CLINICAL TRIAL: NCT03140150
Title: Safety Acceptability and Benefits of Tracking Cardiac Pacemakers by Carelink Express
Acronym: SAFECARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decision by the promoter and funder following recruitment difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: SAFECARE
Record Dates: First submitted 2017-04-13; First posted 2017-05-04 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Telecardiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): A single visit 1 to 3 months after implantation then followed by the attending cardiologist.
  Interventions: Device: Follow-up by Carelink express
- Control Group (Other): A first visit 1 to 3 months after implantation and then every 6 months or every year according to the recommendations of pacemaker follow-up (ie 2 or 4 systematic visits during the follow-up of 2 years).
  Interventions: Other: Follow-up according to the usual recommendations

INTERVENTIONS:
Device: Follow-up by Carelink express — Followed by the cardiologist exclusively using Carelink Express during the study period: a single visit 1 to 3 months after implantation, then followed by the cardiologist and interrogation of the stimulator by Carelink Express
  Arms: Active Group
Other: Follow-up according to the usual recommendations — According to follow-up recommendations for pacemakers, a visit is planned every 6 months if the patient is dependent on the stimulator (either visits to M6, M12, M18 and M24) or annually if the patient is not dependent on the stimulator (visits to M12 and M24).
  Arms: Control Group

SUMMARY:
Follow-up strategy for patients implanted with a pacemaker.

DETAILED DESCRIPTION:
This study seeks to verify that a follow-up strategy for patients implanted with a mono- or double-chamber pacemaker, stimuli-dependent or not, for 2 years, by means of data transmissions of the devices by Carelink Express during the usual consultations with the treating cardiologist significantly reduces the number of unnecessary consultations in the implant centers (without any change in treatment or pacemaker programming) compared to the usual follow-up mode recommended for this type of device.

ELIGIBILITY:
Inclusion Criteria:

* Any patient implanted with a Medtronic brand AAI (R), VVI (R) and DDD (R) cardiac pacemaker, allowing transmission via Carelink Express (Medtronic)
* and accepting inclusion in the study.
* The patient should be followed by a city cardiologist participating in the study.

Exclusion Criteria:

* Age <18 years
* Pregnant or likely to become pregnant during the study
* Patient with an unstable medical condition, NYHA Class IV Heart Failure
* Presence of psychiatric illness, depression, anxiety disorder
* Presence of diseases, other than heart disease, responsible for a reduction in life expectancy for the duration of the study.
* Patient unable to follow protocol (respond to questionnaires)
* Change of residence planned during the study
* Participation in an interventional and therapeutic clinical study; Patient participation in an observational study is permitted.
* Patient not signed consent form
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
At least one unnecessary consultation during two years of follow-up | 2 years
  The primary outcome measure will be at least one unnecessary consultation during two years of follow-up (apart from the first mandatory consultation in all patients)

SECONDARY OUTCOMES:
Occurrence of a serious adverse event | 2 years
  Comparison of the number of serious adverse events during follow-up in each arm (total mortality, hospitalizations for cardiac event, occurrence of a rhythmological event or related to the implanted device)
In-depth sociological study carried out through questionnaires and individual interviews | 2 years
  A more in-depth study will be conducted through questionnaires and individual interviews, developed by sociologists, on representative samples of the two arms of the study (based on age, gender and type of domicile - Individual or collective housing - representative of the populations implanted in 2016) followed at a distance in terms of acceptability, impact on everyday life and the doctor-patient relationship. A survey will also be conducted with attending cardiologists to assess their acceptability of this type of follow-up.
Quality of life | 2 years
  Quality of life questionnaires will be submitted to patients
The medical economic evaluation to measure the efficiency of the device Carelink Express allowing patients' tele-monitoring implanted by a pacemaker | 2 years
  The main analysis will be a comparative cost study based on the following assumption: the direct costs of patient support are different from the direct costs of care for patients undergoing conventional monitoring, in particular in terms of the number Follow-up consultations and transport (COMPAS study: Mabo, 2011).
  The complementary study will be a cost-utility analysis based on a utility measure obtained by the EQ-5D questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mansourati, Professor, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - CHRU Brest, Brest
  - CH Lorient, Lorient